CLINICAL TRIAL: NCT02515383
Title: Preliminary Testing of the MD Anderson Symptom Inventory (Adolescent Version)
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0271; NCI-2020-07335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0271 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Part 1 (MDASI questionnaire, interview): Patients complete the MDASI questionnaire and then complete a cognitive debriefing interview regarding its comprehensibility, the acceptability of each item, and whether any important symptoms are missing from the questionnaire.
  Interventions: Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Part 2 (MDASI questionnaires, interview): Patients complete the MDASI questionnaire twice (1-7 days apart). Approximately 1 week after beginning standard of care treatment, patients complete the MDASI questionnaire at 4 additional time points, each 1 week apart. Patients may also complete a cognitive debriefing interview regarding its comprehensibility, the acceptability of each item, and whether any important symptoms are missing from the questionnaire.
  Interventions: Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Complete cognitive debriefing interview
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete MDASI questionnaire

SUMMARY:
This study investigates how the MD Anderson Symptom Inventory questionnaire modified for use with adolescents performs in adolescent patients with cancer. Conducting interviews with adolescents about the MD Anderson Symptom Inventory may help researchers improve the questionnaire to better understand the symptoms experienced by 13-17 year old patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine how the MD Anderson Symptom Inventory (MDASI) modified for use with adolescents (adolescent version) performs in adolescent patients who have various cancer types, who have undergone various treatments, and who have varying levels of symptom burden.

SECONDARY OBJECTIVES:

I. To explore the feasibility of various methods for collecting MDASI (adolescent version) data (for example, paper-and-pencil forms, face-to-face and telephone interviews, electronic data capture methods such as electronic tablets or automated telephone systems.

II. To evaluate the MDASI (adolescent version) as an estimate of functional status and quality of life in adolescent cancer patients.

OUTLINE:

Part 1: Patients complete the MDASI questionnaire and then complete a cognitive debriefing interview regarding its comprehensibility, the acceptability of each item, and whether any important symptoms are missing from the questionnaire.

Part 2: Patients complete the MDASI questionnaire twice (1-7 days apart). Approximately 1 week after beginning standard of care treatment, patients complete the MDASI questionnaire at 4 additional time points, each 1 week apart. Patients may also complete a cognitive debriefing interview regarding its comprehensibility, the acceptability of each item, and whether any important symptoms are missing from the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and read English
* Diagnosis of cancer, confirmed pathologically or clinically
* Being seen by a healthcare provider at MD Anderson Cancer Center
* Written assent by subject and written consent by parent/guardian for participation
* Starting a cycle of chemotherapy, starting radiation therapy, or starting preparative regimen for stem cell transplantation (Part 2 only)

Exclusion Criteria:

* Medical condition, as determined by the attending physician, that would preclude participation in the study
* Diagnosis of active psychosis, developmental delay, or severe cognitive impairment documented by primary physician in medical record

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents diagnosed with cancer being seen at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance of MD Anderson Symptom Inventory (MDASI) modified for use with adolescents (adolescent version) | Up to 3 months
  Data analysis for the cognitive debriefing portion of the study will be qualitative in nature. Construct validity will be determined using factor analysis. Internal consistency reliability will be assessed using Cronbach coefficient alphas.

SECONDARY OUTCOMES:
Feasibility of collection methods | Up to 3 months
  Patient cognitive debriefing responses about ease of completion based on method and preference for method of completion as well as percentage of successful completions by method during longitudinal assessment in Part 2 will be used to determine the feasibility of the collection methods.
Evaluation of the MDASI (adolescent version) as an estimate of functional status and quality of life | Up to 3 months
  The European Quality of Life Five Dimension Questionnaire (EuroQol EQ-5D) and a single-item quality of life question will be compared to MDASI (adolescent version) symptom severity and interference to establish concurrent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Robert, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org